CLINICAL TRIAL: NCT06487663
Title: Transcatheter Hepatic Artery Chemoembolization Combined With Immune Checkpoint Inhibitors for Liver Tumors
Brief Title: TACE Combined With Immune Checkpoint Inhibitors for Liver Malignant Tumors
Acronym: TIKET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Haipeng Yu, Professor, Tianjin Medical University Cancer Institute and Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCHIO-001
Record Dates: First submitted 2024-06-09; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Cholangiocarcinoma Non-resectable; Liver Metastases; Liver Malignant Tumors
Keywords: Hepatocellular Carcinoma; Cholangiocarcinoma; Liver Metastases; Liver Malignant Tumors
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE combined ICI (Experimental): TACE combined ICI
  Interventions: Procedure: TACE with ICI

INTERVENTIONS:
Procedure: TACE with ICI — Transcatheter hepatic artery chemoembolization and immune checkpoint inhibitors

SUMMARY:
This study will evaluate the efficacy and safety of TACE combined with immune checkpoint inhibitors to treat unresectable hepatocellular carcinoma.

DETAILED DESCRIPTION:
The specific operation of TACE is based on the CSCO Diagnosis and Treatment Guidelines for Primary Liver Cancer (2022 Edition). TACE is performed through microcatheters. After TACE, the coaxial catheter is retained in the hepatic artery or left or right hepatic artery branch. The specific body plan is oxaliplatin+calcium folinate+5-Fu (FOLFOX) (J Hepatol, 2018). Oxaliplatin 85mg/m2 was continuously injected through arterial pump for more than 4 hours on the first day. After HAIC is completed, remove the catheter and sheath. Repeat catheterization in the next treatment cycle.

Immune checkpoint inhibitors can be administered arterial starting after the first TACE treatment, q4w (± 3 days). If the situation requires, the arterial administration of ICI can be adjusted forward or backward for 7 days to adapt to TACE treatment.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of HCC by histology/ cytology or clinical criteria
* Sign informed consent
* When screening for age, the age should be ≥ 18 years old
* Eligible for TACE treatment
* ECOG physical condition score is 0 or 1
* No prior systemic therapy for HCC, especially immunotherapy
* According to the following mRECIST criteria, at least one measurable intrahepatic lesion is suitable for repeated evaluation

Exclusion Criteria:

* Have any history of kidney disease or nephrotic syndrome
* Evidence of extrahepatic spread (EHS)
* Cardiovascular diseases with clinical significance (such as activity), including unstable angina, ≥ grade 2 congestive heart failure, and arrhythmia with poor drug treatment control
* Any condition representing a contraindication to TACE as determined by the investigators
* Known genetic factors for bleeding or thrombosis; Any previous or current evidence indicating a tendency for bleeding
* Individuals who have received immunotherapy (anti PD-1, anti PD-L1, or anti CTLA-4 treatment)
* Previously received HAIC (hepatic artery infusion chemotherapy), TACE (hepatic artery chemoembolization), TAE (hepatic artery embolization), or TARE (hepatic artery radiation embolization)
* Previously received systemic anti-cancer treatment for HCC ,ICC or liver metastasis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2025-10-27 (Estimated); Study Completion 2026-10-27 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 years
  Progression free survival
OS | 3 years
  Overall Survival

SECONDARY OUTCOMES:
ORR | 3 years
  Objective response rate

OTHER OUTCOMES:
TTP | 3 years
  Time to Progression (TTP) as Determined by Investigator
DOR | 3 years
  Duration of Responses (DOR) as Determined by Investigator
AE | Baseline up to approximately 48 months
  Percentage of Participants With Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No